CLINICAL TRIAL: NCT06420622
Title: INDIcators for Clarifying the bAckground of exTreme Obesity in childRen (INDICATOR)
Brief Title: INDIcators for Clarifying the bAckground of exTreme Obesity in childRen
Acronym: INDICATOR
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Antje Koerner, Prof. Dr. med., Prof. Dr. med., University of Leipzig
Other Study IDs: INDICATOR Study
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Gene Abnormality; Child Obesity; Hunger
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples, Whole Exom Sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study investigates the genetic backgrounds of extreme childhood obesity (using saliva sample) and contains short online questionnaires on family history, phenotypical characteristics and hunger behavior. It is an observational study in a predefined cohort (subjects with data in CrescNet aged 0-18 with BMI measurement(s) above the 99.5th percentile). Recruitment will initially be from CrescNet data through the cooperating pediatric and adolescent medical institutions associated with these initiative of data collection in Germany.

DETAILED DESCRIPTION:
In order to be able to investigate the genetic background of extreme obesity, current BMI developments above the 99.5 BMI percentile (extreme obesity) are selected in the existing CrescNet register. Pediatricians (submitting the data) will be informed about these cases. They will be ask to re-identify the patient using the pseudonym (CrescNet-ID) maintained in the registry and to contact the family with a request to participate in the study. The study physician of the study center at the Leipzig University Hospital will take over the study inclusion as well as all necessary clarifications and consents for the study and the genetic examination contained therein. Since the potential probands may live anywhere in Germany, telemedical contact between the study center and the family (interested in participation) will be used.

In addition to the above-mentioned study inclusion, the study physician is also responsible for instructing the family on the correct drawing, collection and sending of saliva samples to the study center, as well as instructing them on how to complete the hyperphagia questionnaire.

At this appointment, the proband is assigned an internal study identification number (INDICATOR-ID). Saliva sample and all questionnaires are assigned to this number.

ELIGIBILITY:
Inclusion Criteria:

* Test subjects older 5 years:

BMI SDS between 0-5 years > 1.881 (= p97) BMI SDS between 5 and 18 >2.567 (=p99.5) Parents and subjects agree that the study information will be provided during a telemedical consultation by the study physician

Exclusion Criteria:

* Known cause of servere early obesity

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cohort from the registry CrescNet (NCT03072537) , data collection of body height and body weight in childhood by primary care pediatricians in Germany
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of each monogenetic obesity | 2 years
  trait among children with early onset severe obesity
Typical patterns of weight gain for each form of obesity | 2 years
  distinguish monogenetic obesity from classical polygenetic forms

SECONDARY OUTCOMES:
Statements about spatial distribution | 2 years
  ZIP-Code related, place of residence of the test subjects
Role of hyperphagia symptoms | 2 years
  method to identify the form of obestity

OTHER OUTCOMES:
Modifying of screening algorithms | 2 Years
  alert pediatricians to a monogenic form of obesity that may be present and treatable

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital University of Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No